CLINICAL TRIAL: NCT07144878
Title: Ultrasonographic Assessment of Parasternal Intercostal Muscle Thickness Versus Rapid Shallow Breathing Index for Predicting Weaning From Mechanical Ventilation
Brief Title: Parasternal Intercostal Ultrasound vs RSBI for Weaning Prediction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Reham Mahmoud Ahmed Shady, Assistant Lecturer of Critical Care Medicine, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD 3-11-2023
Record Dates: First submitted 2025-02-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Insufficiency; Weaning, Ventilator; Respiration, Artificial; Intensive Care Units; Respiratory Muscles
Keywords: Mechanical ventilation; Weaning from ventilation; Extubation outcome; Rapid Shallow Breathing Index (RSBI); Parasternal intercostal muscle ultrasound; Respiratory muscle dysfunction; Spontaneous breathing trial (SBT); Critical care
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: All enrolled patients underwent both RSBI measurement and parasternal intercostal muscle ultrasound prior to spontaneous breathing trial, and outcomes were analyzed by weaning success or failure.
Masking Description: No masking was applied. Both investigators and treating clinicians were aware of the diagnostic tests performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parasternal Intercostal Ultrasound and RSBI Assessment (Other): All enrolled patients underwent ultrasonographic assessment of the parasternal intercostal muscle thickness and calculation of thickening fraction, as well as measurement of the Rapid Shallow Breathing Index (RSBI) using standard ventilator settings. These assessments were performed prior to a 30-minute spontaneous breathing trial. Patients were subsequently classified into successful or failed weaning groups based on trial outcome.
  Interventions: Diagnostic Test: Parasternal Intercostal Ultrasound and RSBI Assessment

INTERVENTIONS:
Diagnostic Test: Parasternal Intercostal Ultrasound and RSBI Assessment — Participants underwent ultrasonographic evaluation of the parasternal intercostal muscle using a high-frequency linear probe to measure thickness and the thickening fraction during respiration. In addition, the Rapid Shallow Breathing Index was calculated from ventilator-displayed values under standardized settings: pressure support equal to zero centimeters of water and positive end-expiratory pressure equal to zero centimeters of water. Both assessments were performed immediately prior to a spontaneous breathing trial to evaluate their predictive accuracy for successful weaning from mechanical ventilation.

SUMMARY:
Mechanical ventilation is essential in the management of critically ill patients, but deciding the proper time to wean and extubate remains a significant challenge. Extubation failure is associated with poor outcomes, including prolonged intensive care unit stay, higher risk of complications, and increased mortality. The rapid shallow breathing index (RSBI) is widely used to predict weaning readiness, but its predictive accuracy is limited. Recently, ultrasound evaluation of respiratory muscles, particularly the parasternal intercostal muscle, has been proposed as a promising bedside tool to assess respiratory effort and load.

This comparative clinical trial was conducted on adult intensive care unit patients at Benha University Hospital who were mechanically ventilated for ≤24 hours and ready for a spontaneous breathing trial. Each patient underwent both rapid shallow breathing index (RSBI) measurement and parasternal intercostal muscle ultrasound prior to the trial. Patients were classified into successful or failed weaning groups based on trial outcome. The study compared the diagnostic accuracy of both methods and aimed to determine whether ultrasound assessment of the parasternal intercostal muscle offers a more reliable predictor of weaning success than rapid shallow breathing index (RSBI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Both sexes
* Patients invasively mechanically ventilated for up to 24 hours and ready to undergo a spontaneous breathing trial
* Patients considered ready for spontaneous breathing trial if all of the following were met:

  * Alert and afebrile
  * Fraction of inspired oxygen less than 50 percent
  * Positive end-expiratory pressure less than or equal to 8 centimeters of water
  * Ratio of arterial oxygen partial pressure to fraction of inspired oxygen greater than 200
  * Arterial blood pH between 7.35 and 7.45
  * Respiratory rate less than or equal to 35 breaths per minute
  * Hemodynamically stable without vasopressor support

Exclusion Criteria:

* Age younger than 18 years
* Pregnancy
* Surgical dressings near or over the sternum that prevent ultrasound examination
* Body mass index less than 18.5 kilograms per square meter (underweight)
* Body mass index greater than or equal to 40 kilograms per square meter (morbid obesity)
* Primary neuromuscular diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of parasternal intercostal muscle thickening fraction measured by ultrasound versus Rapid Shallow Breathing Index for predicting successful weaning from mechanical ventilation | Baseline, immediately prior to the spontaneous breathing trial
  The outcome was assessed by comparing two diagnostic measurements: (1) parasternal intercostal muscle thickening fraction, calculated as the difference between end-inspiratory and end-expiratory muscle thickness divided by end-expiratory thickness, measured using bedside ultrasound; and (2) the Rapid Shallow Breathing Index, calculated as respiratory rate divided by tidal volume, recorded from ventilator-displayed values under standardized zero-support settings. Predictive accuracy for successful weaning was evaluated using receiver operating characteristic analysis, including sensitivity, specificity, positive predictive value, negative predictive value, and area under the curve. Successful weaning was defined as tolerating a 30-minute spontaneous breathing trial without signs of failure.

SECONDARY OUTCOMES:
Sensitivity and specificity of parasternal intercostal muscle thickening fraction and Rapid Shallow Breathing Index in predicting successful weaning | Baseline, immediately prior to the spontaneous breathing trial
  The sensitivity, specificity, positive predictive value, and negative predictive value of parasternal intercostal muscle thickening fraction measured by ultrasound and Rapid Shallow Breathing Index were calculated to assess their ability to predict successful weaning from mechanical ventilation.
Comparison of area under the receiver operating characteristic curve between parasternal intercostal muscle thickening fraction and Rapid Shallow Breathing Index | Baseline, immediately prior to the spontaneous breathing trial
  Receiver operating characteristic curve analysis was performed to compare the diagnostic performance of parasternal intercostal muscle thickening fraction measured by ultrasound and Rapid Shallow Breathing Index. The area under the curve, accuracy, and statistical significance of the difference between the two methods were reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Egypt